CLINICAL TRIAL: NCT00002706
Title: A Phase III Randomized Clinical Trial of Laparoscopic Pelvic and Para-Aortic Node Sampling With Vaginal Hysterectomy and BSO Versus Open Laparotomy With Pelvic and Para-Aortic Node Sampling and Abdominal Hysterectomy and BSO in Endometrial Adenocarcinoma and Uterine Sarcoma, Clinical Stage I, IIA, Grade I, II, III
Brief Title: Laparoscopic Surgery or Standard Surgery in Treating Patients With Endometrial Cancer or Cancer of the Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-LAP2; NCI-2012-02237 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000064513; GOG-LAP2 (Other: Gynecologic Oncology Group); GOG-LAP2 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Endometrial Adenocarcinoma; Stage I Uterine Corpus Cancer; Stage I Uterine Sarcoma; Stage II Uterine Corpus Cancer; Stage II Uterine Sarcoma
MeSH Terms: interventions — Laparoscopy

ARMS (2):
- Arm I (Experimental): Patients undergo vaginal hysterectomy and BSO via laparoscopy.
  Interventions: Procedure: Laparoscopic Surgery; Other: Quality-of-Life Assessment
- Arm II (Active Comparator): Patients undergo total abdominal hysterectomy and BSO via conventional laparotomy.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Laparoscopic Surgery — Undergo vaginal hysterectomy and BSO via laparoscopy
  Other Names: laparoscopic-assisted resection; laparoscopy-assisted surgery
  Arms: Arm I
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo total abdominal hysterectomy and BSO via conventional laparotomy
  Arms: Arm II

SUMMARY:
This randomized phase III trial is studying laparoscopic surgery to see how well it works compared to standard surgery in treating patients with endometrial cancer or cancer of the uterus. Laparoscopic surgery is a less invasive type of surgery for cancer of the uterus and may have fewer side effects and improve recovery. It is not known whether laparoscopic surgery is more effective than standard surgery in treating endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the incidence of surgical complications, peri-operative morbidity, and mortality in patients with stage I or IIa, grade I-III endometrial cancer or uterine cancer undergoing surgical staging through laparoscopic assisted vaginal hysterectomy vs total abdominal hysterectomy.

II. Compare the length of hospital stay after surgery in patients receiving these treatments.

III. Compare the quality of life of patients receiving these treatments. IV. Compare the incidence and location of disease recurrence in patients receiving these treatments.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo vaginal hysterectomy and bilateral salpingo-oophorectomy (BSO) via laparoscopy.

ARM II: Patients undergo total abdominal hysterectomy and BSO via conventional laparotomy.

Patients in both arms also undergo pelvic and para-aortic lymph node sampling. Quality of life is assessed at baseline, at 1, 3, and 6 weeks, and then at 6 months.

Patients are followed at 6 weeks, every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I or IIA, grade I-III endometrial adenocarcinoma or uterine sarcoma
* Must be considered a candidate for surgery
* No contraindication to laparoscopy
* No clinical or chest x-ray evidence of metastasis beyond the uterine corpus or macroscopic involvement of the endocervix
* Performance status - GOG 0-3
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Creatinine no greater than 2.0 mg/dL
* Prior malignancy allowed if no current evidence of disease
* Not pregnant
* No prior pelvic or abdominal radiotherapy
* See Disease Characteristics
* No prior retroperitoneal surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2616 (Actual)
Dates: Start 1996-04; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Duration of disease-free interval | Up to 5 years
  The usual logrank test or a proportional hazards model will be used to assess the equality of the hazard rates between the surgical procedures.
Frequency of aborting LAVH in order to perform an TAH/BSO | Up to 5 years
Frequency of major surgical complications, graded according to the NCI CTC and classified as either less than grade 2 or grade 2 or worse | Up to 5 years
Length of hospitalization following surgery | From the date of surgery to the date of discharge, assessed up to 5 years
  A proportional odds model will be used to estimate the treatment difference while adjusting for potential confounding factors.
Self assessed quality of life scores as measured by FACT-G, Physical Function Subscale from the MOS SF-36, Wisconsin Brief Pain Inventory, Fear of Relapse/Recurrence scale, and Personal Appearance scale | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joan Walker, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bishop EA, Java JJ, Moore KN, Spirtos NM, Pearl ML, Zivanovic O, Kushner DM, Backes F, Hamilton CA, Geller MA, Hurteau J, Mathews C, Wenham RM, Ramirez PT, Zweizig S, Walker JL. Surgical outcomes among elderly women with endometrial cancer treated by laparoscopic hysterectomy: a NRG/Gynecologic Oncology Group study. Am J Obstet Gynecol. 2018 Jan;218(1):109.e1-109.e11. doi: 10.1016/j.ajog.2017.09.026. Epub 2017 Oct 14. PMID 29037481